CLINICAL TRIAL: NCT06474520
Title: An Open Label Clinical Trial to Evaluate the Efficacy and Safety of Calculus Bovis Sativus (CBS) for Idiopathic Inflammatory Demyelinating Disease
Brief Title: Efficacy and Safety of Calculus Bovis Sativus (CBS) for Idiopathic Inflammatory Demyelinating Disease (CBSinIIDD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Jianmin Pharmaceutical Group Co., LTD. (Industry)
Responsible Party: Principal Investigator, Wei Wang, Professor of Neurology, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBSinIIDD
Record Dates: First submitted 2024-06-03; First posted 2024-06-25 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Inflammatory Demyelinating Disease; Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorder; Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease; Acute Disseminated Encephalomyelitis
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Encephalomyelitis, Acute Disseminated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBS therapy, CBS dosage: 100mg per day from day 1 to day 84, in IIDD cohort (Experimental): Subjects in IIDD cohort of this arm will receive general therapy plus CBS.
  Interventions: Drug: Calculus bovis sativus (CBS)
- Control therapy: no intervention, in IIDD cohort. (No Intervention): Subjects in IIDD cohort of this arm will only receive general therapy.
- CBS therapy, CBS dosage: 100mg per day from day 1 to day 84, in healthy cohort (Experimental): Subjects in healthy cohort of this arm will only receive CBS.
  Interventions: Drug: Calculus bovis sativus (CBS)

INTERVENTIONS:
Drug: Calculus bovis sativus (CBS) — Subjects will orally receive 100mg CBS per day from day 1 to day 84.
  Arms: CBS therapy, CBS dosage: 100mg per day from day 1 to day 84, in IIDD cohort; CBS therapy, CBS dosage: 100mg per day from day 1 to day 84, in healthy cohort

SUMMARY:
According to the records of traditional Chinese medicine, CBS has the following functions: clearing the heart, resolving phlegm, promoting bile secretion, and calming the nerves. It can treat fever, coma, delirium, epilepsy, convulsions in children, dental caries, throat swelling, oral sores, carbuncle, and furuncle.

The significant pathophysiological process of primary inflammatory demyelinating disease of the central nervous system (hereinafter referred to as IIDD) is the activation of the immune system of the central nervous system and the enhancement of inflammation. It includes several common diseases: multiple sclerosis (MS), neuromyelitis optica spectrum disorder (NMOSD), myelin oligodendrocyte glycoprotein antibody-related disease (MOGAD), acute disseminated encephalomyelitis (ADEM), concentric sclerosis, tumor-like inflammatory demyelinating disease, etc.

Combined with the inspiration brought to us by the above background research, especially bilirubin and bile acid are closely related to intestinal digestive function, and CBS is clinically effective through oral administration by subjects, the investigators speculate that CBS is likely to exert its immune, anti-inflammatory and neuroprotective effects on the brain by changing the intestinal flora and regulating the brain-gut axis. In terms of symptoms, CBS is likely to have the effect of improving the clinical symptoms of IIDD subjects and reducing disability.

ELIGIBILITY:
Inclusion Criteria:

* IIDD cohort:

  * Subjects are capable of understanding the purpose and risks of the study, providing informed consent and authorizing the use of confidential health information in accordance with national and local privacy regulations.
  * Both men and women are welcome, and the age at the time of providing informed consent is 18-65 years (inclusive).
  * All women of childbearing age and all men must use contraceptive measures during the study and for at least 30 days after the last dose of study treatment. In addition, subjects should not donate sperm or eggs during the study and for at least 30 days after the last dose of study treatment.
  * Must be diagnosed with

    ① Multiple sclerosis, meet the 2017 revised McDonald criteria, and enter the MS cohort;

    ② Aquaporin Protein-4-positive (AQP4) neuromyelitis optica spectrum disease, meet the 2015 international consensus diagnostic criteria for neuromyelitis optica spectrum disease (NMOSD), and AQP4 antibody positive, enter the AQP4-NMOSD cohort;

    ③ Myelin oligodendrocyte glycoprotein antibody-related disease, clinically diagnosed as MOGAD according to the 2023 international MOGAD diagnostic criteria, and positive MOG autoantibody test by cell-based-assay method;

    ④ Acute disseminated encephalomyelitis, clinically diagnosed as ADEM according to the 2013 International Pediatric Multiple Sclerosis Study Group (IPMSSG) diagnostic criteria, characterized by multifocal neurological deficits, must have encephalopathy manifestations (behavioral changes and/or changes in consciousness that cannot be explained by fever, including irritability), and exclude other specific antibody-positive IIDD.
  * EDSS score ≤ 4 points at baseline (visit 1).
  * Stable neurological examination within 30 days prior to Baseline (Visit 1).
* Healthy cohort:

  * Age ≥ 18 years old when signing the informed consent form
  * Healthy adult subjects without underlying diseases

Exclusion Criteria:

* Any clinically significant cardiac, endocrine, hematologic, hepatic, immune, infectious, metabolic, urologic, pulmonary, neurological, dermatologic, psychiatric, and renal disease or other major medical history that the investigator determines would preclude participation in the clinical trial.
* Any untreated teratoma or thymoma at the baseline visit (randomization)
* Other causes of symptoms, including central nervous system infection, septic encephalopathy, metabolic encephalopathy, epileptic disorders, mitochondrial disease, Klein-Levin syndrome, Creutzfeldt-Jakob disease, rheumatic disease, Reyes syndrome, or inborn errors of metabolism.
* History of herpes simplex encephalitis within the previous 24 weeks. 1.5. Any surgical procedure within 4 weeks prior to baseline, except laparoscopic surgery or minor surgery (defined as surgery requiring only local anesthesia or conscious sedation, i.e., surgery that does not require general, neuraxial, or regional anesthesia and can be performed on an outpatient basis; e.g., toenail surgery, mole surgery, wisdom tooth extraction), excluding thymoma or teratoma removal.
* Planned surgery during the study (except minor surgery).
* History of severe allergic or anaphylactic reactions, or any allergic reaction that the investigator believes may be exacerbated by any component of study treatment.
* Current or history of malignant disease, including solid tumors and hematologic malignancies (except for basal cell carcinoma and squamous cell carcinoma that have been completely resected and considered cured for at least 12 months prior to Day -1). Subjects with cancer remission for more than 5 years prior to baseline (Visit 1) may be included after discussion with the sponsor/sponsor approval.
* A history of gastrointestinal surgery (except appendectomy or cholecystectomy performed more than 6 months before screening), irritable bowel syndrome, inflammatory bowel disease (Crohn's disease, ulcerative colitis), or other clinically significant active gastrointestinal diseases in the opinion of the investigator.
* A history of clinically significant recurrent or active gastrointestinal symptoms (e.g., nausea, diarrhea, dyspepsia, constipation) within 90 days before screening, including the need to start symptomatic treatment (e.g., start medication for gastroesophageal reflux disease) or a change in symptomatic treatment within 90 days before screening (e.g., dose increase).
* A history of diverticulitis or concurrent severe gastrointestinal (GI) abnormalities (e.g., symptomatic diverticular disease) because the investigator believes that this may lead to an increased risk of complications such as GI perforation.
* A history of blood donation (1 unit or more), plasma donation, or platelet donation within 90 days before screening.
* Active suicidal ideation within 6 months before screening, or a history of suicide attempt within 3 years before screening.
* Based on the investigator's judgment, there are serious diseases or abnormalities in the clinical laboratory test results that prevent the patient from completing the study or participating in the study safely.
* Pregnant or lactating, or planning to become pregnant during the study or within 3 months after the last dose of the study drug; women of childbearing potential must have a negative serum pregnancy test result at screening and a negative urine pregnancy test result before the start of the study.
* The subject's mental or physical condition will hinder the evaluation of efficacy and safety.
* Systolic blood pressure >150 mmHg or <90 mmHg after sitting still for 5 minutes or before dosing at screening. If out of range, it can be measured again at screening and before dosing. If the repeated measurement value is still out of range, the subject shall not receive the drug.
* Subjects with second or third degree atrioventricular block or sick sinus syndrome, poorly controlled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction, or significant ECG abnormalities, including corrected QT interval >450 msec (male) or 470 msec (female), where corrected QT interval is determined based on the Fridericia correction method, within 3 months prior to the screening visit.
* Planned elective procedures or surgeries at any time after signing the Informed Consent Form by follow-up visit.
* Any condition that affects the absorption of study treatment (e.g., gastrectomy).
* History of hypersensitivity to heparin or history of heparin-induced thrombocytopenia.
* Subjects with abnormalities in medical history, physical examination, ECG, or diagnostic laboratory tests that the investigator considers to be clinically relevant.
* History of human immunodeficiency virus (HIV) or positive test results at screening.
* Current infection with hepatitis C (defined as positive hepatitis C virus (HCV) antibodies and detectable HCV RNA). Subjects with positive HCV antibodies and HCV RNA below the limit of detection are eligible to participate in the study.
* Current infection with hepatitis B (defined as positive HBsAg and/or positive total anti-HBc).
* Chronic, recurrent, or severe infection (e.g., pneumonia, sepsis) within 90 days prior to baseline (visit 1).
* History of tuberculosis (TB) diagnosis or positive latent TB test result.
* Symptoms of bacterial, fungal, or viral infection (including upper respiratory tract infection) within 28 days prior to baseline (visit 1). Subjects with localized fungal infection (e.g., candidiasis, tinea) are eligible for rescreening after successful treatment of the infection.
* Infection requiring hospitalization or IV anti-infective medication within 4 weeks prior to baseline visit.
* Any live or live attenuated vaccine within 28 days prior to baseline (visit 1) or planned during the study.
* Contraindications to all of the following salvage therapies: rituximab, intravenous immunoglobulin, high-dose corticosteroids, or IV cyclophosphamide.
* History of or receipt of the following treatments: Total lymphoid irradiation, cladribine, T-cell or T Cell recipient vaccination, total body irradiation, or total lymphoid irradiation at any time. Stem cell transplantation at any time.
* Abnormal laboratory values determined by the investigator to be clinically significant at Screening or Baseline (Visit 1).
* Any of the following blood test abnormalities at Screening: a. White blood cell count < 3.0 × 10^3/µL. b. Absolute neutrophil count < 2.0 × 10^3/µL. c. Absolute lymphocyte count < 0.5 × 10^3/µL. d. Platelet count < × 10 × 10^4/µL. e. glutamic-pyruvic transaminase, glutamic oxaloacetic transaminase, or γ-glutamyl transpeptidase ≥ 3 x upper limit of normal (ULN) or bilirubin > 2 x ULN. f. glomerular filtration rate ≤ 60 mL/min/1.73 m2. g. Lymphocyte count < lower limit of normal
* Any of the following urine test abnormalities at Screening: a. β-2-microglobulin>0.3 μg/mL. b. Albumin/creatinine ratio>22.6 mg/mmol.
* Previous participation in this study.
* Blood donation (1 unit or more) within 90 days before screening, plasma donation within 1 week before screening, and platelet donation within 6 weeks before screening.
* History of alcohol or drug abuse in the past year (determined by the investigator).
* Pregnant or lactating subjects, as well as subjects planning to become pregnant or start breastfeeding at any time during the study and within 30 days after completion of study treatment.
* Participating in a clinical trial or having participated in a clinical trial within 90 days before screening.
* History of clinically significant suicidal thoughts or behaviors in the past 12 months as assessed by Columbia-Suicide Severity Rating Scale at screening.
* Unwilling or unable to comply with protocol requirements.
* The patient has obvious hearing or vision impairment, language barriers, claustrophobia, etc., which makes the patient unable to cooperate with the neuropsychological scale assessment and MRI examination.
* The researcher or sponsor believes that there are other unknown reasons that make the subject unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The Modified Rankin Scale (mRS) | Up to 12 weeks after treatment initiation
  To assess mRS of subjects within 12 weeks after treatment initiation. The score ranges from 0 to 5. 5 represents the worst.
Expanded Disability Status Scale (EDSS) | Up to 12 weeks after treatment initiation
  To assess EDSS of subjects within 12 weeks after treatment initiation. The score ranges from 0 to 10. 10 represents the worst.
Incidence and Severity of Adverse Effects (AEs) and Severe Adverse Effects (SAEs) | Up to 14 weeks after treatment initiation
  To evaluate the AEs and SAEs occurred within 14 weeks after treatment initiation

SECONDARY OUTCOMES:
The number of newly increased inflammatory lesions on T2 flair weighted imaging at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
The number of newly increased inflammatory lesions on gadolinium-enhanced T1 weighted imaging at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
The score of Mini-mental State Examination (MMSE) at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of MMSE ranges from 0 to 30, and 30 represents the best.
Quantitative and qualitative changes in Montreal cognitive assessment scale (MoCA) at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
The score of Montreal cognitive assessment scale (MoCA) at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of MoCA ranges from 0 to 30, and 30 represents the best.
The score of Hamilton Anxiety Scale at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of Hamilton Anxiety Scale ranges from 0 to 56, and 56 represents the worst.
The score of Hamilton Depression Scale at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of Hamilton Depression Scale ranges from 0 to 81, and 81 represents the worst.
The score of 36-item Short-Form (SF-36) at week 12 compared with baseline (visit 1) and control group. | Up to 12 weeks after treatment initiation
  The score of SF-36 ranges from 0 to 100, and 100 represents the best.
The incidence of Columbia-Suicide Severity Rating Scale (C-SSRS) events at week 14 compared with baseline (visit 1) and control group. | Up to 14 weeks after treatment initiation

OTHER OUTCOMES:
Fecal flora abundance at week 12 compared with baseline (visit 1). | Up to 12 weeks after treatment initiation
Quantitative and qualitative changes in fecal metabolomics analysis at week 12 compared with baseline (visit 1). | Up to 12 weeks after treatment initiation
Profiling of cell subtypes at week 12 compared with baseline (visit 1). | Up to 12 weeks after treatment initiation
The value of SUVmax and ratio of T/B of inflammatory lesion in 18F-DPA-714 PET/MR imaging examinations at week 12 compared with baseline (visit 1). | Up to 12 weeks after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu WJ, Lei T, Yin Z, Pan JH, Chai YS, Xu XY, Yan YX, Wang ZH, Ke J, Wu G, Xu RH, Paranjpe M, Qu L, Nie H. Anti-atherosclerosis and cardio-protective effects of the Angong Niuhuang Pill on a high fat and vitamin D3 induced rodent model of atherosclerosis. J Ethnopharmacol. 2017 Jan 4;195:118-126. doi: 10.1016/j.jep.2016.11.015. Epub 2016 Nov 20. PMID 27880884
- [Background] Zhou J, Jiang T, Wang J, Wu W, Duan X, Jiang H, Jiao Z, Wang X. Multimodal investigation reveals the neuroprotective mechanism of Angong Niuhuang pill for intracerebral hemorrhage: Converging bioinformatics, network pharmacology, and experimental validation. J Ethnopharmacol. 2024 Jan 30;319(Pt 1):117045. doi: 10.1016/j.jep.2023.117045. Epub 2023 Aug 24. PMID 37633621
- [Background] Yu ZJ, Xu Y, Peng W, Liu YJ, Zhang JM, Li JS, Sun T, Wang P. Calculus bovis: A review of the traditional usages, origin, chemistry, pharmacological activities and toxicology. J Ethnopharmacol. 2020 May 23;254:112649. doi: 10.1016/j.jep.2020.112649. Epub 2020 Feb 14. PMID 32068140
- [Background] Shi Y, Xiong J, Sun D, Liu W, Wei F, Ma S, Lin R. Simultaneous quantification of the major bile acids in artificial Calculus bovis by high-performance liquid chromatography with precolumn derivatization and its application in quality control. J Sep Sci. 2015 Aug;38(16):2753-62. doi: 10.1002/jssc.201500139. Epub 2015 Jun 30. PMID 26016891
- [Background] Shimada K, Azuma Y, Kawase M, Takahashi T, Schaffer SW, Takahashi K. Taurine as a marker for the identification of natural Calculus Bovis and its substitutes. Adv Exp Med Biol. 2013;776:141-9. doi: 10.1007/978-1-4614-6093-0_15. PMID 23392879
- [Background] Li X, Yao Y, Chen M, Ding H, Liang C, Lv L, Zhao H, Zhou G, Luo Z, Li Y, Zhang H. Comprehensive evaluation integrating omics strategy and machine learning algorithms for consistency of calculus bovis from different sources. Talanta. 2022 Jan 15;237:122873. doi: 10.1016/j.talanta.2021.122873. Epub 2021 Sep 30. PMID 34736706
- [Background] Liu Y, Tan P, Liu S, Shi H, Feng X, Ma Q. A new method for identification of natural, artificial and in vitro cultured Calculus bovis using high-performance liquid chromatography-mass spectrometry. Pharmacogn Mag. 2015 Apr-Jun;11(42):304-10. doi: 10.4103/0973-1296.153083. PMID 25829769
- [Background] Tang Y, Han Z, Zhang H, Che L, Liao G, Peng J, Lin Y, Wang Y. Characterization of Calculus bovis by principal component analysis assisted qHNMR profiling to distinguish nefarious frauds. J Pharm Biomed Anal. 2023 May 10;228:115320. doi: 10.1016/j.jpba.2023.115320. Epub 2023 Mar 1. PMID 36871364
- [Background] Takahashi K, Azuma Y, Shimada K, Saito T, Kawase M, Schaffer SW. Quality and safety issues related to traditional animal medicine: role of taurine. J Biomed Sci. 2010 Aug 24;17 Suppl 1(Suppl 1):S44. doi: 10.1186/1423-0127-17-S1-S44. PMID 20804621
- [Background] Lu F, Wang L, Chen Y, Zhong X, Huang Z. In vitro cultured calculus bovis attenuates cerebral ischaemia-reperfusion injury by inhibiting neuronal apoptosis and protecting mitochondrial function in rats. J Ethnopharmacol. 2020 Dec 5;263:113168. doi: 10.1016/j.jep.2020.113168. Epub 2020 Jul 27. PMID 32730869
- [Background] Zhong XM, Ren XC, Lou YL, Chen MJ, Li GZ, Gong XY, Huang Z. Effects of in-vitro cultured calculus bovis on learning and memory impairments of hyperlipemia vascular dementia rats. J Ethnopharmacol. 2016 Nov 4;192:390-397. doi: 10.1016/j.jep.2016.09.014. Epub 2016 Sep 9. PMID 27616028
- [Background] Vitek L, Tiribelli C. Bilirubin: The yellow hormone? J Hepatol. 2021 Dec;75(6):1485-1490. doi: 10.1016/j.jhep.2021.06.010. Epub 2021 Jun 18. PMID 34153399
- [Background] Thakkar M, Edelenbos J, Dore S. Bilirubin and Ischemic Stroke: Rendering the Current Paradigm to Better Understand the Protective Effects of Bilirubin. Mol Neurobiol. 2019 Aug;56(8):5483-5496. doi: 10.1007/s12035-018-1440-y. Epub 2019 Jan 5. PMID 30612336
- [Background] Vasavda C, Kothari R, Malla AP, Tokhunts R, Lin A, Ji M, Ricco C, Xu R, Saavedra HG, Sbodio JI, Snowman AM, Albacarys L, Hester L, Sedlak TW, Paul BD, Snyder SH. Bilirubin Links Heme Metabolism to Neuroprotection by Scavenging Superoxide. Cell Chem Biol. 2019 Oct 17;26(10):1450-1460.e7. doi: 10.1016/j.chembiol.2019.07.006. Epub 2019 Jul 25. PMID 31353321
- [Background] Liu HW, Gong LN, Lai K, Yu XF, Liu ZQ, Li MX, Yin XL, Liang M, Shi HS, Jiang LH, Yang W, Shi HB, Wang LY, Yin SK. Bilirubin gates the TRPM2 channel as a direct agonist to exacerbate ischemic brain damage. Neuron. 2023 May 17;111(10):1609-1625.e6. doi: 10.1016/j.neuron.2023.02.022. Epub 2023 Mar 14. PMID 36921602
- [Background] Bhargava P, Smith MD, Mische L, Harrington E, Fitzgerald KC, Martin K, Kim S, Reyes AA, Gonzalez-Cardona J, Volsko C, Tripathi A, Singh S, Varanasi K, Lord HN, Meyers K, Taylor M, Gharagozloo M, Sotirchos ES, Nourbakhsh B, Dutta R, Mowry EM, Waubant E, Calabresi PA. Bile acid metabolism is altered in multiple sclerosis and supplementation ameliorates neuroinflammation. J Clin Invest. 2020 Jul 1;130(7):3467-3482. doi: 10.1172/JCI129401. PMID 32182223
- [Background] Li CX, Wang XQ, Cheng FF, Yan X, Luo J, Wang QG. Hyodeoxycholic acid protects the neurovascular unit against oxygen-glucose deprivation and reoxygenation-induced injury in vitro. Neural Regen Res. 2019 Nov;14(11):1941-1949. doi: 10.4103/1673-5374.259617. PMID 31290452
- [Background] Khalaf K, Tornese P, Cocco A, Albanese A. Tauroursodeoxycholic acid: a potential therapeutic tool in neurodegenerative diseases. Transl Neurodegener. 2022 Jun 4;11(1):33. doi: 10.1186/s40035-022-00307-z. PMID 35659112
- [Background] Hurley MJ, Bates R, Macnaughtan J, Schapira AHV. Bile acids and neurological disease. Pharmacol Ther. 2022 Dec;240:108311. doi: 10.1016/j.pharmthera.2022.108311. Epub 2022 Nov 16. PMID 36400238
- [Background] Jangra A, Gola P, Singh J, Gond P, Ghosh S, Rachamalla M, Dey A, Iqbal D, Kamal M, Sachdeva P, Jha SK, Ojha S, Kumar D, Jha NK, Chopra H, Tan SC. Emergence of taurine as a therapeutic agent for neurological disorders. Neural Regen Res. 2024 Jan;19(1):62-68. doi: 10.4103/1673-5374.374139. PMID 37488845
- [Background] Liu K, Zhu R, Jiang H, Li B, Geng Q, Li Y, Qi J. Taurine inhibits KDM3a production and microglia activation in lipopolysaccharide-treated mice and BV-2 cells. Mol Cell Neurosci. 2022 Sep;122:103759. doi: 10.1016/j.mcn.2022.103759. Epub 2022 Jul 25. PMID 35901929
- [Background] Ohsawa Y, Hagiwara H, Nishimatsu SI, Hirakawa A, Kamimura N, Ohtsubo H, Fukai Y, Murakami T, Koga Y, Goto YI, Ohta S, Sunada Y; KN01 Study Group. Taurine supplementation for prevention of stroke-like episodes in MELAS: a multicentre, open-label, 52-week phase III trial. J Neurol Neurosurg Psychiatry. 2019 May;90(5):529-536. doi: 10.1136/jnnp-2018-317964. Epub 2018 Apr 17. PMID 29666206
- [Background] Martinez-Vacas A, Di Pierdomenico J, Gallego-Ortega A, Valiente-Soriano FJ, Vidal-Sanz M, Picaud S, Villegas-Perez MP, Garcia-Ayuso D. Systemic taurine treatment affords functional and morphological neuroprotection of photoreceptors and restores retinal pigment epithelium function in RCS rats. Redox Biol. 2022 Nov;57:102506. doi: 10.1016/j.redox.2022.102506. Epub 2022 Oct 14. PMID 36270186
- [Background] Zhang F, Deng Y, Wang H, Fu J, Wu G, Duan Z, Zhang X, Cai Y, Zhou H, Yin J, He Y. Gut microbiota-mediated ursodeoxycholic acids regulate the inflammation of microglia through TGR5 signaling after MCAO. Brain Behav Immun. 2024 Jan;115:667-679. doi: 10.1016/j.bbi.2023.11.021. Epub 2023 Nov 19. PMID 37989444